CLINICAL TRIAL: NCT00701012
Title: Comparison of Functional Results of High Ligation and Low Ligation After Anterior Resection for Rectal Cancer - Randomized Controlled Trial-
Brief Title: Comparison of Low and High Ligation in the Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wakayama Medical University (Other)
Responsible Party: Principal Investigator, Hiroki Yamaue, Second Department of Surgery, Wakayama Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WMU512
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Rectal Cancer
Keywords: low or high ligation
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): low ligation, which the IMA is ligated below the origin of the left colic artery
  Interventions: Procedure: preservation of nerve fibers around IMA
- 2 (Active Comparator): high ligation, which the IMA is ligated at its origin from the aorta
  Interventions: Procedure: resection of nerve fibers around IMA

INTERVENTIONS:
Procedure: preservation of nerve fibers around IMA — low ligation
  Other Names: low tie
  Arms: 1
Procedure: resection of nerve fibers around IMA — high ligation
  Other Names: high tie
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the defecatory function when nerve fibers around the inferior mesenteric artery(IMA) and left colic artery(LCA) are preserved(so called low ligation ) or not(high ligation) in the rectosigmoid and rectal cancer surgery.

DETAILED DESCRIPTION:
Fecal incontinence after anterior resection are often observed. Whether or not postoperative bowel function is influenced by the preservation of nerve fibers around the root of IMA and LCA (low ligation) is still unknown. So in this randomized controlled trial, we evaluate the efficacy of low ligation in terms of the bowel function.

ELIGIBILITY:
Inclusion Criteria:

* On the basis of whether anterior resection was anticipated at WMUH for rectosigmoid and rectal cancer, and appropriate informed consent was obtained.

Exclusion Criteria:

* Patients who could not respond to medical interview for own bowel function
* Patients without an informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-01; Primary Completion 2008-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Assessment of bowel function | 1 year

SECONDARY OUTCOMES:
comparison of leakage rate | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hiroki Yamaue, MD, Study Director — Second Departmant of Surgery, Wakayama Medical University
Locations (1):
- Wakayama Medical University, Second Department of Surgery, Kimiidera, Wakayama, Japan

REFERENCES:
- [Background] Uehara K, Yamamoto S, Fujita S, Akasu T, Moriya Y. Impact of upward lymph node dissection on survival rates in advanced lower rectal carcinoma. Dig Surg. 2007;24(5):375-81. doi: 10.1159/000107779. Epub 2007 Aug 4. PMID 17785983
- [Background] Nelson H, Petrelli N, Carlin A, Couture J, Fleshman J, Guillem J, Miedema B, Ota D, Sargent D; National Cancer Institute Expert Panel. Guidelines 2000 for colon and rectal cancer surgery. J Natl Cancer Inst. 2001 Apr 18;93(8):583-96. doi: 10.1093/jnci/93.8.583. PMID 11309435
- [Background] Surtees P, Ritchie JK, Phillips RK. High versus low ligation of the inferior mesenteric artery in rectal cancer. Br J Surg. 1990 Jun;77(6):618-21. doi: 10.1002/bjs.1800770607. PMID 2383724
- [Background] Corder AP, Karanjia ND, Williams JD, Heald RJ. Flush aortic tie versus selective preservation of the ascending left colic artery in low anterior resection for rectal carcinoma. Br J Surg. 1992 Jul;79(7):680-2. doi: 10.1002/bjs.1800790730. PMID 1643485
- [Background] Koda K, Saito N, Seike K, Shimizu K, Kosugi C, Miyazaki M. Denervation of the neorectum as a potential cause of defecatory disorder following low anterior resection for rectal cancer. Dis Colon Rectum. 2005 Feb;48(2):210-7. doi: 10.1007/s10350-004-0814-6. PMID 15711859
- [Background] Iizuka I, Koda K, Seike K, Shimizu K, Takami Y, Fukuda H, Tsuchida D, Oda K, Takiguchi N, Miyazaki M. Defecatory malfunction caused by motility disorder of the neorectum after anterior resection for rectal cancer. Am J Surg. 2004 Aug;188(2):176-80. doi: 10.1016/j.amjsurg.2003.12.064. PMID 15249246
- [Background] Adachi Y, Kakisako K, Sato K, Shiraishi N, Miyahara M, Kitano S. Factors influencing bowel function after low anterior resection and sigmoid colectomy. Hepatogastroenterology. 2000 Jan-Feb;47(31):155-8. PMID 10690600
- [Derived] Matsuda K, Yokoyama S, Hotta T, Takifuji K, Watanabe T, Tamura K, Mitani Y, Iwamoto H, Mizumoto Y, Yamaue H. Oncological Outcomes following Rectal Cancer Surgery with High or Low Ligation of the Inferior Mesenteric Artery. Gastrointest Tumors. 2017 Sep;4(1-2):45-52. doi: 10.1159/000477805. Epub 2017 Jul 5. PMID 29071264
- [Derived] Matsuda K, Hotta T, Takifuji K, Yokoyama S, Oku Y, Watanabe T, Mitani Y, Ieda J, Mizumoto Y, Yamaue H. Randomized clinical trial of defaecatory function after anterior resection for rectal cancer with high versus low ligation of the inferior mesenteric artery. Br J Surg. 2015 Apr;102(5):501-8. doi: 10.1002/bjs.9739. PMID 25764287